CLINICAL TRIAL: NCT03017768
Title: The Effect of Acute Tryptophan Depletion (ATD) on Esophageal Sensitivity in Healthy Volunteers: a Randomized, Single-blind, Placebo-controlled Study
Brief Title: The Effect of Acute Tryptophan Depletion (ATD) on Esophageal Sensitivity in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S57087
Record Dates: First submitted 2016-12-21; First posted 2017-01-11 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2016-12

CONDITIONS: Esophageal Sensitivity
Keywords: Acute tryptophan depletion, esophageal sensitivity,

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute tryptophan depletion (Active Comparator): Administration of an amino acid mixture consisting of 15 amino acids, (4.1g L-alanine, 2.4g glycine, 2.4g L-histidine, 6.0g L-isoleucine, 10.1g L-leucine, 6.7g L-lysine, 4.3g L-phenylalanine, 9.2g L-proline, 5.2g L-serine, 4.3g L-threonine, 5.2g L-tyrosine, 6.7g L-valine, 3.7g L-argine, 2.0g L-cysteine, 3.0g L-methionine) lacking tryptophan to investigate the effect of tryptophan depletion on esophageal sensitivity
  Interventions: Dietary Supplement: Acute tryptophan depletion; Device: Multimodal stimulation probe
- Placebo (Placebo Comparator): Administration of an amino acid mixture consisting of 15 amino acids, (4.1g L-alanine, 2.4g glycine, 2.4g L-histidine, 6.0g L-isoleucine, 10.1g L-leucine, 6.7g L-lysine, 4.3g L-phenylalanine, 9.2g L-proline, 5.2g L-serine, 4.3g L-threonine, 5.2g L-tyrosine, 6.7g L-valine, 3.7g L-argine, 2.0g L-cysteine, 3.0g L-methionine and 3.0g L-trypyophan). Since this amino-acid mixture contains tryptophan it is used as the placebo arm of this cross-over study
  Interventions: Dietary Supplement: Placebo; Device: Multimodal stimulation probe

INTERVENTIONS:
Dietary Supplement: Acute tryptophan depletion — an amino-acid mixture will be administered without tryptophan (active comparator). After an incubation period of 5 hours esophageal sensitivity will be assessed by multimodal stimulation to evaluate the effect of depleted tryptophan levels on esophageal sensitivity
  Arms: Acute tryptophan depletion
Dietary Supplement: Placebo — an amino-acid mixture with tryptophan (placebo mixture) will be administered. After an incubation period of 5 hours esophageal sensitivity will be assessed by multimodal stimulation
  Arms: Placebo
Device: Multimodal stimulation probe — The multimodal esophageal probe allows to perform 4 types of stimulations in the esophagus (thermal, mechanical, electrical and chemical stimulation). These 4 modalities will be evaluated to assess esophageal sensitivity.

SUMMARY:
Esophageal hypersensitivity is considered an important pathophysiological mechanism in patients suffering form non-erosive gastro-esophageal reflux disease. Serotonin (5-HT) is predominantly found in the central nervous system and in the gastro-intestinal (GI) tract. 5-HT plays a major role in the regulation of GI secretion, motility and sensitivity, and has been associated with emotion regulation. Acute tryptophan depletion (ATD) temporarily reduces the availability of tryptophan (TRP), thereby decreasing central and peripheral 5-HT synthesis. From previous studies, ATD is known to affect GI physiology and enhance visceral pain perception in the colon. The aim of the study was to investigate the effect of ATD on esophageal sensitivity in healthy volunteers (HV).

Esophageal multimodal sensitivity was assessed after intragastric infusion of an amino-acid mixture (AA-mix) containing 15 AAs with TRP (control condition) or without TRP (ATD condition). After an incubation period of 5 hours, a probe with a polyurethane bag was positioned in the distal esophagus. Thermal (recirculating a heated saline solution through the bag), mechanical (increasing bag volume), electrical (2 stimulation electrodes) and chemical sensitivity (modified Bernstein) were tested and at 3 time points blood samples were collected for biochemical analysis. General mood was assessed by the Positive and Negative Affect Schedule (PANAS) and the State-Trait Anxiety Inventory (STAI) questionnaires.

DETAILED DESCRIPTION:
1. INTRODUCTION Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. Typical reflux symptoms are heartburn and regurgitation, but GERD can manifest itself through a variety of esophageal and extra-esophageal (atypical) symptoms (e.g. chronic cough).

   In humans, pain is a multimodal experience composed of sensory, physiological and psychological aspects. In order to mimic the clinical situation, experimental models should be based on multimodal testing regimens in which different receptors and central nervous system mechanisms are activated.

   Advances in esophageal sensory stimulation have established that both typical and atypical symptoms may not only arise from acid reflux, but also from reflux events with less acidic pH (pH 4-7). In GERD patients with persisting symptoms in spite of proton pump inhibitor (PPI) treatment (refractory GERD), ongoing weakly acidic reflux is well established as the main underlying factor.

   The basis for symptom generation during weakly-acidic reflux events remains to be elucidated, but acid sensitivity in the pH range 4-7, mechanical distention (enhanced by air in the refluxate), sensitivity to other chemical factors (e.g. bile) and esophageal hypersensitivity to physiological levels of reflux have all been proposed.

   The investigators speculate that visceral hypersensitivity plays an important role in esophageal symptom perception. This is suggested by the reflux parameters that are usual within the physiological number during PPI therapy. Also, previous studies demonstrated that refractory GERD patients on PPI therapy have increased visceral hypersensitivity for thermal, chemical and mechanical esophageal stimulation compared to healthy subjects.

   Serotonin or 5-hydroxytryptamine (5-HT) is a major neurotransmitter predominantly found in the central nervous system and in the gastro-intestinal (GI) tract (mucosal enterochromaffin cells). 5-HT is derived from tryptophan and plays a pivotal role in the regulation of GI secretion, motility and has long been associated with emotion regulation and psychological problems such as depression, anxiety and phobia.

   Acute tryptophan depletion (ATD), which temporarily reduces the availability of the essential amino acid tryptophan (TRP), decreases 5-HT synthesis and is a validated technique to acutely lower central and peripheral 5-HT concentrations. This is accomplished by administration of an amino acid mixture lacking TRP.

   ATD is widely used in psychiatric research to investigate the role of central 5-HT in affective disorders but further research demonstrated that ATD also affects GI physiology by delaying gastric emptying and enhancing visceral pain perception during rectal balloon distention. Furthermore, ATD has been shown to alter gastric postprandial motor function and distension-induced nausea. These findings establish involvement of 5-HT in the control of gastric accommodation and sensitivity.
2. RATIONALE AND OBJECTIVES Multiple studies show that 5-HT is an important player in the brain-gut axis, but its exact role is currently not clear. It was previously shown that acute administration of citalopram, a selective serotonin reuptake inhibitor (SSRI), significantly lowers chemical and mechanical sensitivity in hypersensitive healthy volunteers. Buspirone, a partial 5-HT1A-receptor agonist, is able to modify esophageal motility. The aim of the current study is to investigate the effect of acute tryptophan depletion (ATD) on esophageal sensitivity in a group of healthy volunteers and to evaluate its role in symptom perception.
3. GENERAL DESCRIPTION OF THE STUDY All participants will receive and sign the informed consent before initiation of the study. Esophageal sensitivity will be tested by multimodal stimulation on two sessions (after placebo amino acid solution and after ATD), with an interval of at least one week.
4. MATERIALS AND METHODS Studies will be performed using a multimodal esophageal stimulation probe which allows thermal, mechanical, electrical and chemical stimulations of the esophagus.

During each stimulation, subjects will be instructed to record perception of symptoms using an electronic Visual Analogue Scale (VAS) system. This device allows the subject to scale perception and pain on a scale from 0 to 10.

First perception (VAS=1), pain perception threshold (VAS=5) and pain tolerance threshold (VAS=7) will be recorded. All types of esophageal stimulations will be immediately terminated when the pain tolerance threshold is reached. At the time when the pain tolerance threshold is reached (VAS=7), the subjects will be asked to draw the referred pain area, to identify location and referral area of the pain.

Thermal stimulation will be performed by re-circulating a saline solution (NaCl 0.09%), heated by a water bath, through the balloon mounted on the probe. Stimulation temperature will be steadily increased by increasing the flow rate from the water bath to the balloon. Flow rate will be controlled by a computer operated pump. The volume in the balloon will be kept constant at 5ml to avoid mechanical stimulation of the esophagus. A temperature sensor present in the balloon will continuously monitor the stimulation temperature, which will be displayed online on a computer display throughout the study.

Mechanical stimulation will be performed by distention of the balloon mounted on the probe. The flow of saline (NaCl 0.09%) into the balloon, inducing the distention, is regulated by a computer controlled pump. The volume in the balloon is displayed online on the computer screen throughout the stimulation. Mechanical stimulations will be performed with water of 37°C, to avoid thermal stimulation of the esophagus.

Mechanical stimulation will be preceded by a preconditioning period during which the balloon will be distended until the pain perception threshold (VAS=5) is reached. This preconditioning period is used to precondition the esophageal tissue and to allow the subject to get used to the feeling of mechanical distention.

Electrical stimulation will be performed by 2 stimulation electrodes mounted on proximal to the balloon. Electrical block pulses will be given using a standard electrical stimulator. Single burst pulses will be given with duration of 1ms at 200Hz.The amplitude of the pulses will steadily increase, with steps of 0.5mA and an interval of 15 seconds. For safety, the maximum intensity is limited to 50 mA. ECG monitoring will be performed as a safety measure during the electrical stimulations of the esophagus.

Chemical stimulation will be performed in the distal esophagus by infusing an acidic solution (HCl 0.1N) in the esophagus. Infusion rate is controlled by a peristaltic infusion pump with a flow rate of 2ml/min. The stimulation will last for a maximum of 30 minutes.

Acute tryptophan depletion

The effect of ATD on esophageal sensitivity will be studied. The amino acid mixture will be prepared according to a protocol previously used by the investigators. All substrates are commercially available with an isotopic and chemical purity of minimal 99%. The identity of the products will be confirmed using gas chromatography - mass spectrometry (GC-MS, GC-column: AT5-MS 30m x 0.25 mm iternal diameter; 0.25µm film (Grace)). The amino acid mixture consists of 15 amino acids, (4.1g L-alanine, 2.4g glycine, 2.4g L-histidine, 6.0g L-isoleucine, 10.1g L-leucine, 6.7g L-lysine, 4.3g L-phenylalanine, 9.2g L-proline, 5.2g L-serine, 4.3g L-threonine, 5.2g L-tyrosine, 6.7g L-valine, 3.7g L-argine, 2.0g L-cysteine, 3.0g L-methionine and 3.0g L-trypyophan). The TRP-deficient amino acid mixture consists of the same 15 amino acids but lacking tryptophan.

The amino acid mixture will be administered via a nasogastric probe to avoid nausea due to the unpleasant taste and smell of the mixture. During placebo sessions, a control amino acid mixture is used, containing the same amino acids enriched with TRP in order to prevent a decrease in TRP levels. Over time, each participant will receive placebo or ATD in the first session in a random sequence. In the second session, the subject will receive the other product that he/she didn't receive the first time. Because the amino acid mixture will influence the levels of 5-HT of the HV we will first exert the Mini International Neuropsychiatric Interview (dutch, version 5.0.0, DSM-IV) during the recruitment of the volunteers to evaluate their psychiatric condition.

STUDY OUTLINE After an overnight fast subjects will come to the endoscopy unit of the UZ Gasthuisberg, where the study will be performed. Two sessions will be scheduled for every subject: one placebo and one ATD session, with at least one week interval between each of the sessions. Sessions will run in a single-blind way, the order of placebo and ATD will be randomized.

Since maximal TRP depletion is obtained approximately 5 hours after intake of the amino acid mixture, the amino acid will be administered through nasogastric infusion 5 hours prior to the actual start of the esophageal stimulations.

During the time between administration of the amino acid mixture and the actual start of esophageal stimulations, the subjects will be asked to watch standardized movies with a neutral emotional content. Five hours after the administration of the amino acid mixture, the multimodal stimulation probe will be positioned through the mouth. After the probe is positioned in the esophagus (10 cm above the lower esophageal sphincter), it will be fixed to the chin and the subject will remain in in semi-recumbent position for the entire study period. Before the start of the stimulations, there will be an adaptation period of 15 minutes for the subjects, to get used to the feeling of the probe and to provide instructions for the correct use of the VAS meter.

VAS scores will be monitored during each type of stimulation. All stimulations will be immediately stopped at the moment the subject reaches the pain tolerance threshold (VAS=7) except for the electrical stimulation, where we will stop the stimulation after reaching VAS 5, for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

- Age between 18 and 60 years old

Exclusion Criteria:

* history of psychiatric disease or a positive first degree psychiatric family history,
* pregnancy or lactation,
* concomitant administration of any centrally activating medication
* medication affecting esophageal motility,
* significant co-morbidities (neuromuscular, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic),
* prior history of esophageal, Ear-Nose and Throat or gastric surgery or endoscopic anti-reflux procedure,
* history of gastrointestinal disease
* During the last two weeks before the study, the volunteers should be free from medication, except for oral contraceptives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Measurement of changes in esophageal sensitivity after acute tryptophan depletion assessed by multimodal esophageal stimulation protocol | 2 sessions per HV with at least one week interval, duration of each session: approximately 7 hours. Temperature stimulation: 30 minutes
  Investigation of the effect of acute tryptophan depletion on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the Temperature values (°C) of the stimulation tests between the placebo and acute tryptophan depletion condition to see if tryptophan depletion affects the sensitivity to increasing temperature.
Measurement of changes in esophageal sensitivity after acute tryptophan depletion | 2 sessions per HV with at least one week interval, duration of each session: approximately 7 hours. Mechanical stimulation: 30 minutes
  Investigation of the effect of acute tryptophan depletion on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the balloon volumes (volume in ml) of the stimulation tests between the placebo and acute tryptophan depletion condition to see if tryptophan depletion affects the sensitivity to increasing balloon volume.
Measurement of changes in esophageal sensitivity after acute tryptophan depletion | 2 sessions per HV with at least one week interval, duration of each session: approximately 7 hours. Electrical stimulation: 30 minutes
  Investigation of the effect of acute tryptophan depletion on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the tolerated intensity of the electrical pulses (mA) of the stimulation tests between the placebo and acute tryptophan depletion condition to see if tryptophan depletion affects the sensitivity to increasing electrical pulses.
Measurement of changes in esophageal sensitivity after acute tryptophan depletion | 2 sessions per HV with at least one week interval, duration of each session: approximately 7 hours. Chemical stimulation: 30 minutes
  Investigation of the effect of acute tryptophan depletion on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the volume of infused acid (ml) of the stimulation tests between the placebo and acute tryptophan depletion condition to see if tryptophan depletion affects the sensitivity to acid infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, M.D., PhD, Principal Investigator — TARGID, KU Leuven
Locations (1):
- Targid, KU Leuven, Leuven, Vlaams-Brabant, Belgium